CLINICAL TRIAL: NCT04332523
Title: A Single-Dose, Open-Label, Parallel-Group Study to Evaluate the Effect of Mild, Moderate, and Severe Hepatic Impairment on the Pharmacokinetics of JNJ-53718678
Brief Title: A Study of JNJ-53718678 in Participants With Hepatic Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A strategic decision was made to discontinue the study. The decision was not based on a safety concern.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108773; 53718678RSV1010 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-04-01; First posted 2020-04-02 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — JNJ-53718678

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Participants with Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment will receive a single oral dose of JNJ-53718678 suspension on Day 1.
  Interventions: Drug: JNJ-53718678
- Group 2: Participants with Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment will receive a single oral dose of JNJ-53718678 suspension on Day 1.
  Interventions: Drug: JNJ-53718678
- Group 3: Participants with Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment will receive a single oral dose of JNJ-53718678 suspension on Day 1.
  Interventions: Drug: JNJ-53718678
- Group 4: Participants with Normal Hepatic Function (Experimental): Participants with normal hepatic function will receive a single oral dose of JNJ-53718678 suspension on Day 1.
  Interventions: Drug: JNJ-53718678

INTERVENTIONS:
Drug: JNJ-53718678 — Participants will receive a single oral dose of JNJ-53718678 suspension on Day 1.
  Other Names: Rilematovir

SUMMARY:
The main purpose of the study is to evaluate the pharmacokinetc (PK) of a single oral dose of JNJ-53718678 in participants with varying degrees of impaired hepatic function (mild, moderate, and severe) when compared with participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* A woman of childbearing potential must have a negative serum (beta human chorionic gonadotropin [beta-HCG]) test at screening and on Day -1 of the treatment period
* Contraceptive use by female participants or women should be consistent with local regulations regarding the use of contraceptive methods for participant participating in clinical studies
* If a woman, must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 30 days after receiving the study drug
* A male participant must agree not to donate sperm for the purpose of reproduction from Day -1 of the study and for a minimum of 90 days after receiving the study drug
* For participants with mild, moderate or severe hepatic impairment: the participants must have a total Child-Pugh score of 5 to 6, inclusive (mild); or 7 to 9, inclusive (moderate); or 10-15, inclusive (severe). The Investigator will determine degree of hepatic impairment

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to JNJ-53718678 or its excipients
* Donated blood or blood products or had substantial loss of blood (more than 500 milliliter [mL]) within 90 days before the administration of study drug or intention to donate blood or blood products during the study
* Received an experimental drug (including investigational vaccines) or used an experimental medical device within 30 days or within a period less than 5 times the drug's half-life, whichever is longer, before the dose of the study drug is scheduled
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments
* Preplanned surgery or procedures that would interfere with the conduct of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of JNJ-53718678 | Predose, 15 minutes (min), 30 min, 1 hour (h), 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 16h, 24h, 36h, 48h, 72h and 96h postdose
  Cmax is defined as the maximum plasma concentration of JNJ-53718678.
Area Under the Plasma Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration (AUClast) of JNJ-53718678 | Predose, 15 min, 30 min, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 16h, 24h, 36h, 48h, 72h and 96h postdose
  AUClast is defined as the area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration of JNJ-53718678.
Area Under the Plasma Concentration-time Curve From Time 0 to Infinite Time (AUC[0-infinity]) | Predose, 15 min, 30 min, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 16h, 24h, 36h, 48h, 72h and 96h postdose
  AUC(0-infinity) is defined as the area under the plasma concentration-time curve from time 0 to infinite time calculated as the sum of AUClast and Clast/lz, in which Clast is the last observed quantifiable concentration.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | From screening up to Day 14 (Up to 42 days)
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - The Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency